CLINICAL TRIAL: NCT04351724
Title: A Multicenter, Randomized, Active Controlled, Open Label, Platform Trial on the Efficacy and Safety of Experimental Therapeutics for Patients With COVID-19 (Caused by Infection With Severe Acute Respiratory Syndrome Coronavirus-2)
Brief Title: Austrian CoronaVirus Adaptive Clinical Trial (COVID-19)
Acronym: ACOVACT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Kaiser Franz Josef Hospital (Other); SMZ-Ost Donauspital (Other); Otto Wagner Hospital (Other); Hospital Hietzing (Other); Wilhelminenspital Vienna (Other); Medical University Innsbruck (Other); Medical University of Graz (Other); Kepler University Hospital (Other)
Responsible Party: Principal Investigator, Bernd Jilma, Univ.Prof.Dr. Bernd Jilma, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACOVACT
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Chloroquine; Hydroxychloroquine; Lopinavir; Rivaroxaban; candesartan; remdesivir; pentaglobulin

STUDY DESIGN:
Intervention Model Description: Three main study arms (antiviral treatments) and three substudies (A, B, C) are planned. The main study arms are exclusive, while patients from the main study arms may participate in one or more substudies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- (Hydroxy)Chloroquine (STOPPED) (Experimental): Due to limited availability of the experimental substances, this arm will include both chloroquine and hydroxychloroquine treatment. However, both substances are similar chemically and also with regards to the mechanism of action comparable.
  Dosage: Hydroxychloroquine 200mg 2-0-2 on day 1 followed by 200mg 1-0-1, or Chloroquine 250mg 2-0-2, as available
  Interventions: Drug: Chloroquine or Hydroxychloroquine
- Lopinavir/Ritonavir (Experimental): Dosage: 200mg/50mg 4-0-4 on day 1 and 3-0-3 thereafter
  Interventions: Drug: Lopinavir/Ritonavir
- Standard of Care (Other): patients will be treated with "standard of care", which precludes treatment with lopinavir/ritonavir or (hydroxy-)chloroquine
  Interventions: Other: Best standard of care
- Rivaroxaban (Experimental): 5mg 1-0-1
  Interventions: Drug: Rivaroxaban
- Thromboprophylaxis (Active Comparator): according to local standard
  Interventions: Drug: Thromboprophylaxis
- RAS Blockade (Experimental): Renin-Angiotensin-System-Blockade (RAS) by candesartan intake starting with 4mg once daily and titrated to normotension patients > 120/80 mmHG are eligible
  Interventions: Drug: Candesartan
- non-RAS-Blockade (Active Comparator): non-RAS blocking antihypertensive agents titrated to normotension Those with normal blood pressure may only be controlled without further treatment
  Interventions: Drug: non-RAS blocking antihypertensives
- Asunercept 25mg (Experimental): 25mg 1x per week, maximum of four doses only patients with oxygen requirement
  Interventions: Drug: Asunercept 25mg
- Asunercept 100mg (Experimental): 100mg 1x per week, maximum of four doses only patients with oxygen requirement
  Interventions: Drug: Asunercept 100mg
- Asunercept 400mg (Experimental): 400mg 1x per week, maximum of four doses only patients with oxygen requirement
  Interventions: Drug: Asunercept 400mg
- Best Standard of Care - Control Group for Asunercept (Other): only patients with oxygen requirement
  Interventions: Other: Best standard of care
- Remdesivir (Experimental): 200mg loading dose on day 1, 100mg for a total treatment duration of 5-10 days
  Interventions: Drug: Remdesivir
- Pentaglobin (Experimental): Patients treated at the intensive care unit only, continuous infusion of 7ml/kg/day over 12h for 5 days
  Interventions: Drug: Pentaglobin
- best standard of care (Other): Patients treated at the intensive care unit only
  Interventions: Other: Best standard of care

INTERVENTIONS:
Drug: Chloroquine or Hydroxychloroquine — Hydroxychloroquine 200mg 2-0-2 on day 1 followed by 200mg 1-0-1, or Chloroquine 250mg 2-0-2, as available
  Arms: (Hydroxy)Chloroquine (STOPPED)
Drug: Lopinavir/Ritonavir — Lopinavir/Ritonavir 200mg/50mg 2-0-2
  Arms: Lopinavir/Ritonavir
Other: Best standard of care — best standard of care
  Arms: Best Standard of Care - Control Group for Asunercept; Standard of Care; best standard of care
Drug: Rivaroxaban — 2.5mg 2-0-2 or 10mg 1/2-0-1/2, as applicable
  Arms: Rivaroxaban
Drug: Thromboprophylaxis — as local standard, most likely to be low molecular weight heparin
  Arms: Thromboprophylaxis
Drug: Candesartan — starting dose 4mg once daily, titrated to normotension
  Arms: RAS Blockade
Drug: non-RAS blocking antihypertensives — This excludes angiotensin converting enzyme inhibitors (ACEi) and angiotensin receptor blockers (AT-blockers, sartans) and includes alpha-receptor antagonists, calcium antagonists, amongst others
  Arms: non-RAS-Blockade
Drug: Remdesivir — 200mg on day 1, thereafter 100mg for a total of 5-10 treatment days, according to local standards
  Arms: Remdesivir
Drug: Asunercept 400mg — asunercept 400mg once per week, up to 4 doses in total
  Arms: Asunercept 400mg
Drug: Asunercept 100mg — asunercept 100mg once per week, up to 4 doses in total
  Arms: Asunercept 100mg
Drug: Asunercept 25mg — asunercept 25mg once per week, up to 4 doses in total
  Arms: Asunercept 25mg
Drug: Pentaglobin — 7ml/kg/day for 12h for 5 days
  Arms: Pentaglobin

SUMMARY:
The Austrian Coronavirus Adaptive Clinical Trial (ACOVACT) is a randomized, controlled, multicenter, open-label basket trial that aims to compare various antiviral treatments for COVID-19. Moreover three substudies have been integrated. Currently, patients will be randomized to receive (hydroxy-)chloroquine (Treatment stopped after reports of safety issues), lopinavir/ritonavir, remdesivir or standard of care. Moreover, these patients are eligible for substudy A (randomized to rivaroxaban 5mg 1-0-1 vs. standard of care), substudy B (renin-angiotensin (RAS) blockade vs. no RAS blockade for patients with blood pressure >120/80mmHg), and substudy C (asunercept vs standard of care, pentglobin vs. standard of care for patients with respiratory deterioration and high inflammatory biomarkers).

Endpoints were chosen based on the master protocol published by the World Health Organisation and include a 7-point scale of clinical performance, mortality, oxygen requirement (both dose and type), duration of hospitalization, viral load and safety.

ELIGIBILITY:
Inclusion Criteria

Laboratory confirmed (i.e. PCR-based assay) infection with SARS-CoV-2 (ideally but not necessarily

≤72 hours before randomization for "antiviral" treatments) OR radiological signs of COVID-19 in chest X-ray or computed tomography

* Hospitalisation due to SARS-CoV-2 infection, except for sub-study B, which may also include outpatients with COVID-19
* Requirement of oxygen support (due to oxygen saturation <94% on ambient air or >3% drop in case of chronic obstructive lung disease)
* Informed Consent obtained, the patient understands and agrees to comply with the planned study procedures, except for sub-study C: obtaining informed consent may be impossible due to the severe condition of the patient and may be waived
* ≥18 years of age
* Sub-study A: not on chronic anticoagulation Sub-study B: Sub-study B: blood pressure ≥130/85mmHg in 2 consecutive measurements OR patients with established and treated hypertension
* Sub-study B: Control group 1: Patients with suspicion of but negative tests for COVID-19. This group may consist of hospitalized and non-hospitalized patients.
* Sub-study B: healthy volunteers
* Sub-study C: Signs of respiratory deterioration and progressing inflammation: need for oxygen supplementation, non-invasive ventilation, high-flow oxygen devices or mechanical ventilation AND CRP levels >5mg/dL (for Pentaglobin only) and ICU admission (for Pentaglobin only)
* For female patients with childbearing potential: willingness to perform effective measures of contraception during the study

Exclusion Criteria

* Moribund, or estimated life expectancy <1 month (e.g. terminal cancer, etc.)
* Patient does not qualify for intensive care, based on local triage criteria
* Pregnancy or breastfeeding
* Severe liver dysfunction (e.g. ALT/AST > 5 times upper limit of normal)
* Stage 4 chronic kidney disease or requiring dialysis for direct anticoagulant treatment
* Allergy or intolerances to experimental substance (ineligibility for treatment arm), for Asunercept known hereditary fructose intolerance
* Anticipated discharge from hospital within 48 hours (for any given reason)
* Contraindications for treatment arm 2 (lopinavir/ritonavir): severe hepatic impairment, CYP3A4/5 metabolized drugs, as deemed relevant by treating physicians
* Contraindications for treatment arm 3 (remdesivir): <40kg bodyweight
* Known active HIV or viral hepatitis
* Substudy A contraindications for rivaroxaban: active bleeding or bleeding diathesis, lesion or condition considered as major risk factor for bleeding, recent brain or spinal injury, recent brain or spinal or ophthalmic surgery, recent intracranial hemorrhage, known or suspected esophageal varices, arteriovenous malformations, vascular aneurysms, major intraspinal or intracerebral vascular abnormalities, ongoing therapeutic anticoagulation, which will be continued, according to clinical practice
* Sub-study B contraindications for nitrendipine: chronic heart failure, allergies, hypersensitivities and intolerances, severe hepatic impairment and/or cholestasis, concomitant therapy with aliskirencontaining medications (for patients with diabetes mellitus or a GFR<60ml/min/1.73m2), known significant bilateral renal artery stenosis or renal artery stenosis of a solitary kidney
* Sub-study C contraindications for IL-6 blockade: Contraindications: allergies and intolerances, active untreated diverticulitis, inflammatory bowel disease, any treatment with an IL-6 or IL-6R blocking drug (e.g. tocilizumab, sarilumab, siltuximab) <30 days before study inclusion.
* Sub-study C: Known active tuberculosis.
* Asunercept: females of childbearing potential
* Sub-study C with Pentaglobin: Contraindications to Pentaglobin

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
sustained improvement (>48h) of one point on the WHO Scale | Inclusion to day 29, daily evaluation
  The primary endpoint is time to clinical improvement which is defined as time from randomization to an (sustained) improvement of at least one category on two consecutive days compared to the status at randomization measured on a seven-category ordinal scale (proposed by WHO).
  The 7-categories of the World Health Organization proposed scale, as follows:
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or ECMO;
  7. Death.
  During hospitalization this score will be determined daily (till day 29). If a patient is released from the hospital before day 29, the score will be determined at day 11 and 29 after randomization (depending when the patient was released or by telephone call).

SECONDARY OUTCOMES:
Time to improvement on WHO Scale | Inclusion to day 29, daily evaluation
  The scale described in the primary endpoint is used
Mean change in the ranking on an ordinal scale from baseline | Inclusion to day 29, daily evaluation
  The scale described in the primary endpoint is used
time to discharge or a National Early Warning Score (NEWS) ≤2 (maintained for 24h), whichever occurs first | Inclusion to day 29, daily evaluation
  the National Early Warning Score includes respiratory rate, oxygen saturation, use of supplemental oxygen, temperature, systolic blood pressure, heart rate and levels of consciousness (AVPU Scale)
change from baseline in National Early Warning Score (NEWS) | Inclusion to day 29, daily evaluation
  The scale described in the primary endpoint is used
Oxygenation free days | Inclusion to day 29, daily evaluation
Incidence of new oxygen use during the trial | Inclusion to day 29, daily evaluation
  new oxygen may include insufflation or oxygen mask, high flow oxygen devices, non-invasive ventilation devices or mechanical ventilation
duration of oxygen use during the trial | Inclusion to day 29, daily evaluation
Ventilator free days until day 29 | Inclusion to day 29, daily evaluation
  number of days with requirement of mechanical ventilation
Incidence of new mechanical ventilation use during the trial | Inclusion to day 29, daily evaluation
duration of mechanical ventilation use during the trial | Inclusion to day 29, daily evaluation
Viral load/viral clearance | Inclusion to day 29, daily evaluation
  obtained by polymerase chain reaction in nasal/oropharyngeal swabs, performed at baseline and then three times a week, if possible
Duration of Hospitalization | Inclusion to day 29, daily evaluation
Mortality | 15-day, 29-day, 60-day, 90-day mortality
Obesity - mortality | BMI at admission, mortality until day 29
  BMI (kg/m2), within all subjects the impact of obesity on overall mortality will be investigated
Obesity - duration of hospitalization | BMI at admission, duration of hospitalization until day 29 or discharge
  BMI (kg/m2) , within all subjects the impact of obesity on the duration of hospitalization will be investigated
Obesity - ICU admission | BMI at admission, ICU admission until day 29 or discharge
  BMI (kg/m2) , within all subjects the impact of obesity on ICU admission will be investigated
Obesity - new oxygen use | BMI at admission, new oxygen use until day 29 or discharge
  BMI (kg/m2) new oxygen may include insufflation or oxygen mask, high flow oxygen devices, non-invasive ventilation devices or mechanical ventilation
Drug-drug interactions with lopinavir/ritonavir | Inclusion to day 29, daily evaluation
  lopinavir and ritonavir both interact with numerous other drugs by inhibiting the cytochrome enzymes 3A4. Using commercially available drug-interaction programs, the number and severity grading of drug-drug-interactions will be documented (for instance uptodate interaction tool, medscape). This is an exploratory analysis of drug-drug interactions with the above mentioned substances. severity grading usually encompass "contraindicated", "serious", "monitor closely", "minor" interaction.
Renin Angiotensin System (RAS) fingerprint | Inclusion to day 29, daily evaluation
  for sub-study B only: RAS fingerprint measures metabolites involved in the renin-angiotensin-system. The influence of randomized treatment with candesartan (RAS blockade) will be analyzed
SpO2/FiO2 ratio | Inclusion to day 29, daily evaluation
  for sub-study C only
paO/FiO2 ratio | Inclusion to day 29, daily evaluation
  for sub-study C only, for ICU patients only
modified Sequential Organ Failure Assessment | Inclusion to day 29, daily evaluation
  for sub-study C only
C-reactive protein | baseline, day 2, 3, 4, 5, 7
  unit mg/dL
Interleukin-6 | baseline, day 2, 3, 4, 5, 7
  unit pg/mL
procalcitonin | baseline, day 2, 3, 4, 5, 7
  unit ng/mL
IgM Concentrations | baseline, day 2, 3, 4, 5, 7
  unit mg/dL
IgA Concentrations | baseline, day 2, 3, 4, 5, 7
  unit mg/dL
differential blood counts | baseline, day 2, 3, 4, 5, 7

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Jilma, MD, Principal Investigator — Medical University of Vienna
Locations (9):
- Austria (9):
  - Medical University of Innsbruck, Innsbruck, Tyrol
  - Medical University of Graz, Graz
  - Kepler University Hospital, Linz
  - Medical University of Vienna, Vienna
  - Wilhelminenspital, Vienna
  - SMZ Süd Kaiser Franz Josef Spital, Vienna
  - KH Hietzing, Vienna
  - SMZ Baumgartner Höhe Otto Wagner Spital, Vienna
  - SMZ Ost Donauspital, Vienna

IPD SHARING:
Plan to Share IPD: No
Anonymized and pseudonymized data will be published in peer reviewed journals and may be presented at congresses and conferences

REFERENCES:
- [Derived] Gleiss A. Visualizing a marker's degrees of necessity and of sufficiency in the predictiveness curve. BMC Med Res Methodol. 2025 Apr 23;25(1):107. doi: 10.1186/s12874-025-02544-y. PMID 40269760
- [Derived] Hofstetter L, Tinhof V, Mayfurth H, Kurnikowski A, Rathkolb V, Reindl-Schwaighofer R, Traugott M, Omid S, Zoufaly A, Tong A, Kropiunigg U, Hecking M. Experiences and challenges faced by patients with COVID-19 who were hospitalised and participated in a randomised controlled trial: a qualitative study. BMJ Open. 2022 Oct 11;12(10):e062176. doi: 10.1136/bmjopen-2022-062176. PMID 36220325
- [Derived] Karolyi M, Pawelka E, Omid S, Koenig F, Kauer V, Rumpf B, Hoepler W, Kuran A, Laferl H, Seitz T, Traugott M, Rathkolb V, Mueller M, Abrahamowicz A, Schoergenhofer C, Hecking M, Assinger A, Wenisch C, Zeitlinger M, Jilma B, Zoufaly A. Camostat Mesylate Versus Lopinavir/Ritonavir in Hospitalized Patients With COVID-19-Results From a Randomized, Controlled, Open Label, Platform Trial (ACOVACT). Front Pharmacol. 2022 Jul 22;13:870493. doi: 10.3389/fphar.2022.870493. eCollection 2022. PMID 35935856
- [Derived] Heber S, Pereyra D, Schrottmaier WC, Kammerer K, Santol J, Rumpf B, Pawelka E, Hanna M, Scholz A, Liu M, Hell A, Heiplik K, Lickefett B, Havervall S, Traugott MT, Neubock MJ, Schorgenhofer C, Seitz T, Firbas C, Karolyi M, Weiss G, Jilma B, Thalin C, Bellmann-Weiler R, Salzer HJF, Szepannek G, Fischer MJM, Zoufaly A, Gleiss A, Assinger A. A Model Predicting Mortality of Hospitalized Covid-19 Patients Four Days After Admission: Development, Internal and Temporal-External Validation. Front Cell Infect Microbiol. 2022 Jan 24;11:795026. doi: 10.3389/fcimb.2021.795026. eCollection 2021. PMID 35141170
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343